CLINICAL TRIAL: NCT04122703
Title: A Randomized Controlled Trial Investigating the Efficacy of Percutaneous Tibial Nerve Stimulation (PTNS) in the Treatment of Female Sexual Dysfunction (FSD)
Brief Title: Trial of Tibial Nerve Stimulation for Treating Sexual Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jason Kim, Clinical Assistant Professor of Urology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1370654
Record Dates: First submitted 2019-10-06; First posted 2019-10-10 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Female Sexual Dysfunction
Keywords: Percutaneous Tibial Nerve Stimulation; Female Sexual Dysfunction; Sexual dysfunction; peripheral neuromodulation
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: We will be recruiting 66 patients, who will be randomized (1:1) to either the PTNS group or the Sham group.
Who Masked: Participant, Care Provider
Masking Description: Patients in both PTNS and Sham groups will come to the clinic once a week for 30 sessions, and will not know their group assignment until the end of the study.
  All the interventions will be performed by the sub-investigator. The care providing physician will not know the group assignment of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Percutaneous tibial nerve stimulation (PTNS) (Experimental): The patients in the PTNS group will receive 1 PTNS treatments per week for 12 weeks.
  Interventions: Device: percutaneous tibial nerve stimulation (PTNS)
- Transcutaneous electrical nerve stimulation (TENS) (Sham Comparator): The patients in the Sham group will receive one sham (TENS) treatment per week for 12 weeks
  Interventions: Device: Sham procedure

INTERVENTIONS:
Device: percutaneous tibial nerve stimulation (PTNS) — The PTNS treatments will be given in 30 min sessions. The PTNS treatment consists of inserting a 34-gauge needle electrode approximately 5 cm cephalad to the medial malleolus and, as well as placing a PTNS surface electrode on the ipsilateral calcaneus. To keep the electrode placement consistent with the sham treatment, 2 inactive transcutaneous electrical nerve stimulation (TENS) surface electrodes are also added, 1 placed under the little toe and 1 on the top of the foot. The PTNS lead set is connected to the Urgent PC stimulator, and a current level of 0.5 to 10 mA at 20 Hz is delivered until the flexion of the big toe is observed or the patient reports a radiating sensation at the sole of the foot.
  Arms: Percutaneous tibial nerve stimulation (PTNS)
Device: Sham procedure — The sham treatment, involves simulating the sensation of the PTNS needle insertion at the same location using a Steritberger placebo needle. This is a blunt tip needle which simulates the sensation of a needle prick when touched to the skin, however, the blunt tip retracts into the handle when pressed into the skin. This creates the illusion of the needle entering the skin, without breaking the skin's surface. An inactive PTNS surface electrode is also placed on the ipsilateral calcaneus. The two TENS surface electrodes, placed in the same location as the PTNS treatment, are active and deliver stimulation mimicking the sensory effects of the PTNS. However, since no electrode needles were inserted near the tibial nerve, there will be no tibial nerve stimulation
  Arms: Transcutaneous electrical nerve stimulation (TENS)

SUMMARY:
The purpose of this study is to understand the efficacy of PTNS versus a placebo in the treatment of female sexual dysfunction syndrome.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the efficacy of PTNS in treating patients with FSD. We will be recruiting 66 patients, who will be randomized (1:1) to either the PTNS group or the Sham group. The patients in the PTNS group will receive one PTNS treatment per week for 12 weeks. The patients in the Sham group will receive one sham treatment per week for 12 weeks. Patients in both groups will be asked to complete questionnaires before the start of the treatment, as well as after 12-weeks of treatment to assess the changes in the severity of their symptoms

Aim 1: To evaluate the effect of percutaneous tibial nerve stimulation (PTNS), compared to a validated sham, on sexual functioning in women with female sexual dysfunction (FSD).

Aim 2: To compare the effect of PTNS on lower urinary tract symptoms versus sexual functioning in patient with FSD.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or older
* FSFI score of ≤ 26.55
* Patients must be sexually active within one month prior to the study and plans to continue to be sexually active for the next 12 weeks (Sexual activity can include masturbating, vaginal intercourse, caressing, and foreplay)

Exclusion Criteria:

* Patients with anatomical limitations preventing successful placement of the electrode (bleeding disorders, peripheral vascular disease, ulcers, or lower leg cellulitis)
* Patients with medical disorders precluding stimulation (cardiac pacemakers, current use of Holter monitor, known history of neuropathy)
* Pregnant women or women intending to become pregnant during the course of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Female Sexual Function Index (FSFI) | Baseline, at week 6 and at week 12
  Female Sexual Function Index (FSFI) is a 19-item questionnaire used to assess female sexual function. Minimum score is 1.2 and maximum score is 36. A score of 26.55 or lower is classified as sexual dysfunction

SECONDARY OUTCOMES:
Change in Arizona Sexual Experiences Scale (ASEX) | Baseline, at week 6 and at week 12
  Arizona Sexual Experiences Scale (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Possible total scores range from 5 to 30, with the higher scores indicating more sexual dysfunction.
Change in Prolapse/Urinary Incontinence Sexual-12 (PISQ-12 ) Function Questionnaire (PISQ- 12) | Baseline, at week 6 and at week 12
  PISQ-12 is a 12-item questionnaire used to assess sexual function in women with pelvic organ prolapse or urinary incontinence. Possible total scores range from 0 to 48, with the lower scores indicating more sexual dysfunction.
Change in Urinary Distress Inventory (UDI-6) | Baseline, at week 6 and at week 12
  Urinary Distress Inventory (UDI-6) is a 6-item questionnaire used to assess lower urinary tract symptoms in women. Possible total scores range from 0 to 18, with the higher scores indicating more urogenital distress.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Kim, MD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook Medicine Women's Pelvic Health And Continence Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters KM, Carrico DJ, Perez-Marrero RA, Khan AU, Wooldridge LS, Davis GL, Macdiarmid SA. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. J Urol. 2010 Apr;183(4):1438-43. doi: 10.1016/j.juro.2009.12.036. Epub 2010 Feb 20. PMID 20171677
- [Background] Zimmerman LL, Gupta P, O'Gara F, Langhals NB, Berger MB, Bruns TM. Transcutaneous Electrical Nerve Stimulation to Improve Female Sexual Dysfunction Symptoms: A Pilot Study. Neuromodulation. 2018 Oct;21(7):707-713. doi: 10.1111/ner.12846. Epub 2018 Sep 3. PMID 30247794